CLINICAL TRIAL: NCT03748953
Title: China Continuation: A Single-Arm, Open-Label Study of Oral Ixazomib Maintenance Therapy After Initial Therapy in Patients With Newly Diagnosed Multiple Myeloma Not Treated With Stem Cell Transplantation
Brief Title: Study of Oral Ixazomib Maintenance Therapy After Initial Therapy in Participants With Newly Diagnosed Multiple Myeloma Not Treated With Stem Cell Transplantation (SCT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C16021 CCS; 2014-001394-13 (EudraCT Number); NCT04371770 (obsolete NCT alias)
Record Dates: First submitted 2018-11-16; First posted 2018-11-21 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
Keywords: Drug Therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ixazomib (Experimental): Participants received ixazomib 3 milligrams (mg), capsules, orally, once on Days 1, 8, and 15 for Cycles 1 through 4, during which if the participants tolerated the initial dose, the dose was escalated to ixazomib 4 mg, capsules, orally, once on Days 1, 8, and 15 for Cycles 5 through 26, or until documented PD or intolerable toxicity, whichever occurred first (cycle length=28 days).
  Interventions: Drug: Ixazomib

INTERVENTIONS:
Drug: Ixazomib — Ixazomib Capsules

SUMMARY:
The purpose of this study is to determine the long-term safety and tolerability of ixazomib maintenance therapy.

DETAILED DESCRIPTION:
The drug being tested in this study is called ixazomib. Ixazomib is being tested to slow disease progression and improve overall survival in Chinese participants who have newly diagnosed multiple myeloma (NDMM) who have had a major positive response to initial therapy and have not undergone stem cell transplantation (SCT). This study will look at the effect of ixazomib has on the length of time that participants are free of disease progression and their overall survival. After the implementation of Amendment 8, participants who received placebo-matching capsules before unblinding and have not yet experienced disease progression will cross over to receive ixazomib.

The study will enroll approximately 37 patients. Participants will be assigned to a single treatment group

• Ixazomib

All participants will be asked to take one capsule on Days 1, 8, and 15 of every 28-day cycle, for up to approximately 24 months (equivalent to 26 cycles [if no cycle delays], to the nearest complete cycle) or until documented progressive disease (PD) or intolerable toxicity, whichever occurs first.

This multi-center trial will be conducted in China. The overall time to participate in this study is until a total of approximately up to 60 months. Participants will make multiple visits to the clinic, and every 4 weeks until the next line of therapy begins for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female participants aged 18 years or older with a confirmed diagnosis of symptomatic NDMM according to standard criteria.
2. Has completed 6 to 12 months (±2 weeks) of initial therapy, during which the participant was treated to best response, defined as the best response maintained for 2 cycles after the M-protein nadir is reached.
3. Has documented major response (partial response [PR], very good partial response [VGPR], complete response [CR]) according to the international myeloma working group (IMWG) uniform response criteria, version 2011, after this initial therapy.
4. Female participants who:

   Are postmenopausal for at least 1 year before the screening visit, OR Are surgically sterile, OR If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 90 days after the last dose of study drug, or Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [e.g., calendar, ovulation,symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)

   Male participants, even if surgically sterilized (i.e., status postvasectomy), who:

   Agree to practice effective barrier contraception during the entire study Treatment period and through 90 days after the last dose of study drug, or Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal are not acceptable methods of contraception.)
5. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
6. Has availability of complete documentation for:

   1. Details of initial disease state, initial therapy, and response
   2. Cytogenetic assessment at diagnosis (cytogenetic assessment performed after diagnosis must be approved by a Takeda project clinician or designee)
   3. International Staging System (ISS) staging at diagnosis (requiring beta 2-microglobulin and serum albumin results).
7. Has Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2.
8. Suitable venous access for the study-required blood sampling and consent for the specific amounts that will be taken.
9. Participant is willing and able to adhere to the study visit schedule and other protocol requirements including blood sampling and bone marrow aspiration.
10. Participants must meet the following clinical laboratory criteria at study entry:

1. Absolute neutrophil count (ANC) ≥1,000/mm^3 without growth factor support and platelet count ≥ 75,000/mm^3. Platelet transfusions to help participants meet eligibility criteria are not allowed within 3 days before enrollment.

2. Total bilirubin ≤1.5*the upper limit of the normal range (ULN). 3. Alanine aminotransferase and aspartate aminotransferase ≤3*ULN. 4. Calculated creatinine clearance ≥30 mL/min (using the Cockroft-Gault equation).

Exclusion Criteria:

1. Has multiple myeloma that relapsed after, or was not responsive to, initial therapy.
2. Had prior stem-cell transplantation (SCT).
3. Has radiotherapy within 14 days before enrollment.
4. Had been diagnosed or treated for another malignancy within 5 years before enrollment or previously diagnosed with another malignancy with evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
5. Female participants who are lactating and breastfeeding or have a positive serum pregnancy test during the Screening period.
6. Has major surgery within 14 days before enrollment.
7. Has central nervous system involvement.
8. Infection requiring intravenous (IV) antibiotic therapy or other serious infection within 14 days before enrollment.
9. Has diagnosis of Waldenstrom's macroglobulinemia, polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome, plasma cell leukemia, primary amyloidosis, myelodysplastic syndrome, or myeloproliferative syndrome.
10. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, uncontrolled congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
11. Systemic treatment with strong cytochrome P450 (CYP3A) inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital) or use of St. John's wort within 14 days before enrollment.
12. Ongoing or active infection, known human immunodeficiency virus positive, active hepatitis B or C infection.
13. Has comorbid systemic illnesses or other severe concurrent disease that, in the judgment of the investigator, would make the participant inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens (e.g., peripheral neuropathy (PN) that is Grade 1 with pain or Grade 2 or higher of any cause).
14. Psychiatric illness/social situation that would limit compliance with study requirements.
15. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
16. Inability to swallow oral medication, inability or unwillingness to comply with the drug administration requirements, or gastrointestinal (GI) procedure that could interfere with the oral absorption or tolerance of treatment.
17. Treatment with any investigational products within 30 days before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (10):
- China (10):
  - Beijing Chaoyang Hospital Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital (the First Affiliated Hospital With Nanjing Medical University), Nanjing, Jiangsu
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Chang Zheng Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - 1st Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b603a4db2bf003ab4a2b7?idFilter=%5B%22C16021CSC%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 37 participants (31 enrolled in this study and 6 rolled over from study C16021[NCT02312258]) with a diagnosis of newly diagnosed multiple myeloma (NDMM) not treated with stem cell transplantation (SCT) took part in the study at investigative sites in China from 24 January 2019 to 06 December 2023.
Pre-assignment Details: Of the 31 participants who newly enrolled in this study, 10 (4 randomized to placebo and 6 to ixazomib) were enrolled before the implementation of Protocol Amendment 08, and 21 under the amendment, with all 21 receiving ixazomib as the study design was changed to a single-arm study. After Amendment 08, 2 of the 4 participants who were initially randomized to placebo crossed over to the ixazomib arm. As per planned analysis, these 4 participants were not included in the Efficacy Population.
Groups:
- Ixazomib: Participants received ixazomib 3 mg, capsules, orally, once on Days 1, 8, and 15 for Cycles 1 through 4, during which if the participants tolerated the initial dose, the dose was escalated to ixazomib 4 mg, capsules, orally, once on Days 1, 8, and 15 for Cycles 5 through 26, or until documented progressive disease (PD) or intolerable toxicity, whichever occurred first (cycle length=28 days).
- Placebo: Participants received ixazomib placebo-matching capsules, orally, once on Days 1, 8, and 15 of each cycle until Protocol Amendment 08 was implemented (cycle length=28 days).
Period: Treatment Prior to Amendment 08
Arm/Group | Ixazomib | Placebo
Started | 6 | 4
Placebo Safety Population (Placebo Safety Population included all participants who received at least 1 dose of placebo.) | 0 | 4
Completed | 6 | 0
Not Completed | 0 | 4
Not completed — Discontinued to Switch to Ixazomib | 0 | 2
Not completed — Reason not Specified | 0 | 2
Period: Treatment Post Amendment 08
Arm/Group | Ixazomib | Placebo
Started | 35 (6 participants (initially receiving ixazomib, before Protocol Amendment 08 was implemented) continued to receive ixazomib after implementation of Amendment 08 and 2 participants who received placebo before Amendment 08 switched to ixazomib after the implementation.) | 0
Efficacy Population (Efficacy Population included all participants who received ixazomib treatment for the duration of their study participation. Participants who were randomized to the placebo arm and crossed over to the ixazomib arm upon implementation of Amendment 08 were not included.) | 33 | 0
Ixazomib Safety Population (Ixazomib Safety Population included all participants who received at least 1 dose of ixazomib.) | 35 | 0
Completed | 0 | 0
Not Completed | 35 | 0
Not completed — Withdrawal by Subject | 18 | 0
Not completed — Reason not Specified | 16 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Efficacy Population included all participants who received ixazomib treatment for the duration of their study participation. As prespecified in the statistical analysis plan (SAP), the Efficacy Population contained only one arm i.e., Ixazomib (data for the participants who received placebo before Protocol Amendment 8 was not collected per statistical analysis plan), thus data is presented accordingly.
Arm/Group | Ixazomib
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.80 (7.551)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 33
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Categorized According to Performance Status (PS) Based on Eastern Cooperative Oncology Group (ECOG) PS
Description: ECOG PS was used to assess physical health of participants. ECOG PS grade:0= fully active, able to carry on all pre-disease performance without restriction,1= restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature 2= ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours, 3= capable of only limited self-care, 4= completely disabled, cannot carry on any selfcare, totally confined to bed or chair confined to bed or chair more than 50% of waking hours and 5= dead. Only those categories with non-zero values were reported.
Time Frame: Month 25
Population: Ixazomib Safety Population (ISP) included all participants who received at least 1 dose of ixazomib. As prespecified in the SAP, the ISP contained only one arm i.e., Ixazomib (participants originally randomized to ixazomib + participants who were randomized to the placebo arm prior to implementation of Amendment 08 and who crossed over to ixazomib arm contributing data for this outcome measure from the time they initiated ixazomib onward), thus data is presented accordingly.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib
Number analyzed (Participants) | 35
Participants
  ECOG Score 0 | 34
  ECOG Score 1 | 1

2. Primary Outcome: Percentage of Participants Receiving Ixazomib With Treatment-emergent Adverse Events (TEAEs)
Description: Adverse events (AEs) were defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through 30 days after the last dose of study drug. A TEAE was defined as an AE that started or worsened after first study drug administration and within 30 days of last dose of study drug. Percentages are rounded off to the nearest whole number.
Time Frame: Up to 58.4 months
Population: ISP included all participants who received at least 1 dose of ixazomib. As prespecified in the SAP, the ISP contained only one arm i.e., Ixazomib (participants originally randomized to ixazomib + participants who were randomized to the placebo arm prior to implementation of Amendment 08 and who crossed over to ixazomib arm contributing data for this outcome measure from the time they initiated ixazomib onward), thus data is presented accordingly.
Measure: Number; unit: percentage of participants
Arm/Group | Ixazomib
Number analyzed (Participants) | 35
percentage of participants | 97

3. Primary Outcome: Percentage of Participants Receiving Ixazomib With Treatment-emergent Serious Adverse Events (SAEs)
Description: AEs were defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through 30 days after the last dose of study drug. A TEAE was defined as an AE that started or worsened after first study drug administration and within 30 days of last dose of study drug. An SAE was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability or incapacity, was a congenital abnormality or birth defect, or is an important medical event. Percentages are rounded off to the nearest whole number.
Time Frame: Up to 58.4 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Ixazomib
Number analyzed (Participants) | 35
percentage of participants | 31

4. Primary Outcome: Number of Participants Receiving Ixazomib With Clinically Significant Changes in Safety Laboratory Values
Description: Clinical laboratory assessments included hematology, serum chemistry, and urinalysis. Any clinically significant changes in the clinical laboratory value over time based on the investigator's interpretation were reported.
Time Frame: Up to 58.4 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib
Number analyzed (Participants) | 35
Participants | 0

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the date of first dose of study drug to the first occurrence of PD as evaluated by the investigator or death from any cause, whichever occurred first. PD was defined as ≥25% increase from lowest value in serum M component or urine M-component; difference between involved and uninvolved free light chain (FLC) levels (absolute increase >10 milligrams per deciliter [mg/dL]); bone marrow plasma cell percent ≥10%; new bone lesions or soft tissue plasmacytomas development or definite increase in existing bone lesions/soft tissue plasmacytomas size; hypercalcaemia development.
Time Frame: From the first dose of study drug to every 4 weeks until PD or death from any cause (up to 58.4 months)
Population: Efficacy Population included all participants who received ixazomib treatment for the duration of their study participation. As prespecified in the SAP, the Efficacy Population contained only one arm i.e., Ixazomib (efficacy outcomes data for the participants who received placebo before Protocol Amendment 8 was not collected per statistical analysis plan), thus data is presented accordingly.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib
Number analyzed (Participants) | 33
months | 21.3 [9.20 to NA] — Upper limit of 95% confidence interval (CI) was not estimable due to censoring.

6. Secondary Outcome: Overall Survival (OS)
Description: OS was measured as the time from the date of first dose of study drug to the date of death.
Time Frame: From the first dose of study drug to every 12 weeks during follow-up after PD or next line therapy or death whichever occurred later (up to 58.4 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib
Number analyzed (Participants) | 33
months | NA [NA to NA] — Median, lower limit, and upper limit of 95% CI were not estimable due to censoring.

7. Secondary Outcome: Percentage of Participants Who Achieved or Maintained Best Response Before PD or up to Subsequent Therapy
Description: Response was assessed according to International Myeloma Working Group (IMWG) criteria. Best response includes partial response (PR), very good partial response (VGPR), and complete response (CR). PR as per IMWG criteria is 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to less than (<)200 mg per 24 hours. VGPR is serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein plus urine M-protein level <100 mg per 24 hours. CR is negative immunofixation of serum and urine and disappearance of soft tissue plasmacytomas and <5% plasma cells in bone marrow. Percentages are rounded off to the nearest whole number.
Time Frame: Up to 58.4 months
Population: Response-evaluable Population included a subset of the Efficacy Population and consisted of all participants who had a baseline&at least 1 postbaseline response assessment. As prespecified in the SAP, this population contained only one arm i.e., Ixazomib (efficacy outcomes data for the participants who received placebo before Protocol Amendment 8 was not collected per SAP), thus data is presented accordingly.
Measure: Number; unit: percentage of participants
Arm/Group | Ixazomib
Number analyzed (Participants) | 33
percentage of participants
  PR | 3
  VGPR | 12
  CR | 76

8. Secondary Outcome: Duration of Complete Response (CR)
Description: Duration of CR was defined as the time from the date of first dose of study drug or the date of CR to the date of first documentation of PD. CR was defined as negative immunofixation on the serum and urine; soft tissue plasmacytomas disappearance; <5% plasma cells (PCs) in bone marrow.
Time Frame: Up to 58.4 months
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib
Number analyzed (Participants) | 33
months | NA [12.88 to NA] — Median and upper limit of 95% CI were not estimable due to censoring.

9. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from the date of first dose of study drug to the date of first documentation of PD. PD was defined as ≥25% increase from lowest value in serum M component or urine M-component; difference between involved and uninvolved FLC levels (absolute increase >10 mg/dL); bone marrow plasma cell percent ≥10%; new bone lesions or soft tissue plasmacytomas development or definite increase in existing bone lesions/soft tissue plasmacytomas size; hypercalcaemia development.
Time Frame: Up to 58.4 months
Population: Efficacy Population included all participants who received ixazomib treatment for the duration of their study participation. As prespecified in the SAP, the Efficacy Population contained only one arm i.e., Ixazomib (efficacy outcomes data for the participants who received placebo before Protocol Amendment 8 was not collected per SAP), thus data is presented accordingly.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib
Number analyzed (Participants) | 33
months | 21.3 [9.20 to NA] — Upper limit of 95% CI was not estimable due to censoring.

10. Secondary Outcome: Time to Next-Line Therapy (TTNT)
Description: TTNT was defined as the time from the date of first dose of study drug to the date of the first dose of next-line of antineoplastic therapy.
Time Frame: Up to 58.4 months
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib
Number analyzed (Participants) | 33
months | NA [24.48 to NA] — Median and upper limit of 95% CI were not estimable due to censoring.

11. Secondary Outcome: Percentage of Participants With A New Primary Malignancy
Time Frame: Up to 58.4 months
Population: ISP=all participants who received atleast 1 dose of ixazomib. As prespecified in SAP,ISP had only 1 arm:Ixazomib (participants originally randomized to ixazomib + participants randomized to placebo arm prior to implementation of Amendment 08 & crossed over to ixazomib arm contributing data for this OM from time they initiated ixazomib onward), thus data is presented accordingly.
Measure: Number; unit: percentage of participants
Arm/Group | Ixazomib
Number analyzed (Participants) | 35
percentage of participants | 0

12. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 as Measured by the Global Health Status (GHS)
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. The change from baseline in GHS (EORTC QLQ-C30) score is presented. Participant responses to the question "How would you rate your overall health during the past week?" are scored on a 7-point scale (1=very poor to 7=excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall GHS.
Time Frame: Baseline, Cycle 26 (cycle length=28 days)
Population: Efficacy Population included all participants who received ixazomib treatment for the duration of their study participation. Overall number of participants analyzed is the number of participants with data available for analyses. As prespecified in the SAP, the Efficacy Population contained only one arm i.e., Ixazomib (efficacy outcomes data for the participants who received placebo before Protocol Amendment 8 was not collected per SAP), thus data is presented accordingly.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixazomib
Number analyzed (Participants) | 11
score on a scale | -5.3 (15.49)

13. Secondary Outcome: Correlation Between Frailty Status and PFS
Description: Participant's frailty status is classified as fit, unfit, or frail on the basis of 4 components: age, the Charlson comorbidity scoring system without age weighting, the Katz index of independence in activities of daily living, and the Lawton instrumental activities of daily living scale. The sum of the 4 frailty scores equals the total frailty score. A total frailty score of 0 corresponds to a frailty status of fit; a total score of 1, to unfit; and a total score of 2 or more, to frail. PFS is defined as the time from the date of first dose of study drug to the first occurrence of PD as evaluated by the investigator.
Time Frame: Up to 58.4 months
Population: Efficacy Population included all participants who received ixazomib treatment for the duration of their study participation. Number analyzed is the number of participants with data available for analysis for the specified category. As prespecified in the SAP, the Efficacy Population contained only one arm i.e., Ixazomib (efficacy outcomes data for the participants who received placebo before Protocol Amendment 8 was not collected per SAP), thus data is presented accordingly.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib
Number analyzed (Participants) | 33
months
  Frailty Status: Fit: number analyzed (Participants) | 25
  Frailty Status: Fit | NA [12.68 to NA] — Median and upper limit of 95% CI were not estimable due to censoring.
  Frailty Status: Unfit: number analyzed (Participants) | 5
  Frailty Status: Unfit | 20.9 [0.89 to NA] — Upper limit of 95% CI was not estimable due to censoring.
  Frailty Status: Frail: number analyzed (Participants) | 3
  Frailty Status: Frail | 6.5 [6.18 to NA] — Upper limit of 95% CI was not estimable due to censoring.

14. Secondary Outcome: Correlation Between Frailty Status and OS
Description: Participant's frailty status is classified as fit, unfit, or frail on the basis of 4 components: age, the Charlson comorbidity scoring system without age weighting, the Katz index of independence in activities of daily living, and the Lawton instrumental activities of daily living scale. The sum of the 4 frailty scores equals the total frailty score. A total frailty score of 0 corresponds to a frailty status of fit; a total score of 1, to unfit; and a total score of 2 or more, to frail. OS was measured as the time from the date of first dose of study drug to the date of death.
Time Frame: Up to 58.4 months
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib
Number analyzed (Participants) | 33
months
  Frailty Status: Fit: number analyzed (Participants) | 25
  Frailty Status: Fit | NA [NA to NA] — Median, lower limit, and upper limit of 95% CI were not estimable due to censoring.
  Frailty Status: Unfit: number analyzed (Participants) | 5
  Frailty Status: Unfit | NA [NA to NA] — Median, lower limit, and upper limit of 95% CI were not estimable due to censoring.
  Frailty Status: Frail: number analyzed (Participants) | 3
  Frailty Status: Frail | NA [NA to NA] — Median, lower limit, and upper limit of 95% CI were not estimable due to censoring.

15. Secondary Outcome: Plasma Concentration of Ixazomib
Description: Plasma concentrations of the complete hydrolysis product of ixazomib citrate (ixazomib) were measured using a validated liquid chromatography-tandem mass spectrometry (LC/MS/MS) assay.
Time Frame: Cycle 1 (1 and 4 hours post-dose Day 1, Days 8 and 15 pre-dose); Cycle 2 and 5 (Days 1 and 8 pre-dose) and Cycles 3, 4, 6 to 10 (Day 1 pre-dose) (cycle length=28 days)
Population: ISP=all participants who received atleast 1 dose of ixazomib. Number analyzed=participants with data available for analysis at specified time point. As prespecified in SAP, ISP had only 1 arm:Ixazomib (participants originally randomized to ixazomib + participants randomized to placebo arm prior to implementation of Amendment 08 & crossed over to ixazomib arm contributing data for this OM from time they initiated ixazomib onward), thus data is presented accordingly.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Ixazomib
Number analyzed (Participants) | 35
nanograms per milliliter (ng/mL)
  Cycle 1 Day 1: 1 Hour Post-dose | 15.3 (181)
  Cycle 1 Day 1: 4 Hours Post-dose | 16.6 (94.4)
  Cycle 1 Day 8: Pre-dose: number analyzed (Participants) | 34
  Cycle 1 Day 8: Pre-dose | 2.25 (51.5)
  Cycle 1 Day 15: Pre-dose | 4 (53.6)
  Cycle 2 Day 1: Pre-dose | 2.92 (46.8)
  Cycle 2 Day 8: Pre-dose: number analyzed (Participants) | 34
  Cycle 2 Day 8: Pre-dose | 4.37 (42.5)
  Cycle 3 Day 1: Pre-dose: number analyzed (Participants) | 34
  Cycle 3 Day 1: Pre-dose | 3.15 (41.9)
  Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 31
  Cycle 4 Day 1: Pre-dose | 3.16 (59.4)
  Cycle 5 Day 1: Pre-dose: number analyzed (Participants) | 29
  Cycle 5 Day 1: Pre-dose | 3.25 (42.1)
  Cycle 5 Day 8: Pre-dose: number analyzed (Participants) | 21
  Cycle 5 Day 8: Pre-dose | 5.29 (36.9)
  Cycle 6 Day 1: Pre-dose: number analyzed (Participants) | 29
  Cycle 6 Day 1: Pre-dose | 3.58 (41.3)
  Cycle 7 Day 1: Pre-dose: number analyzed (Participants) | 28
  Cycle 7 Day 1: Pre-dose | 4.04 (48.5)
  Cycle 8 Day 1: Pre-dose: number analyzed (Participants) | 23
  Cycle 8 Day 1: Pre-dose | 3.28 (64.7)
  Cycle 9 Day 1: Pre-dose: number analyzed (Participants) | 19
  Cycle 9 Day 1: Pre-dose | 3.7 (31.3)
  Cycle 10 Day 1: Pre-dose: number analyzed (Participants) | 19
  Cycle 10 Day 1: Pre-dose | 2.99 (37.6)

16. Secondary Outcome: Time to Resolution of Peripheral Neuropathy (PN) Events
Description: PN is defined as the event in the high-level term of peripheral neuropathies not elsewhere classified (NEC) according to the medical dictionary for regulatory activities (MedDRA). A PN event was considered as resolved if its final outcome was resolved with no subsequent PN event of the same preferred term occurring on the resolution date or the day before and after. Time to resolution was defined as the time from the initial onset date (inclusive) to the resolution date for resolved events.
Time Frame: Up to 58.4 months
Population: ISP=all participants who received atleast 1 dose of ixazomib. Overall number of participants analyzed=participants with PN events. As prespecified in SAP,ISP had only 1 arm:Ixazomib (participants originally randomized to ixazomib+participants randomized to placebo prior to Amendment 08 &crossed over to ixazomib arm contributing data for this OM from time they initiated ixazomib onward),& is presented accordingly.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ixazomib
Number analyzed (Participants) | 3
days | 24.0 [7.0 to NA] — Upper limit of 95% CI was not estimable due to censoring.

17. Secondary Outcome: Time to Improvement of PN Events
Description: PN is defined as the event in the high-level term of peripheral neuropathies NEC according to the MedDRA. A PN event is considered to be improved if the event improves from the maximum grade; that is, all the grades recorded after the maximum grade are less than the maximum grade. Time to improvement is defined as the time from the initial onset date (inclusive) of the maximum grade to the first onset date that the toxicity grade is below the maximum grade with no higher grade thereafter, or the resolution date, whichever occurs first.
Time Frame: Up to 58.4 months
Population: ISP=all participants who received atleast 1 dose of ixazomib. Overall number of participants analyzed=participants with PN events. As prespecified in SAP,ISP had only 1 arm:Ixazomib (participants originally randomized to ixazomib + participants randomized to placebo arm prior to implementation of Amendment 08 & crossed over to ixazomib arm contributing data for this OM from time they initiated ixazomib onward), thus data is presented accordingly.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ixazomib
Number analyzed (Participants) | 3
days | 8.0 [7.0 to NA] — Upper limit of 95% CI was not estimable due to censoring.

ADVERSE EVENTS:
Time Frame: Up to 58.4 months
Description: Ixazomib Safety Population included all participants who received at least 1 dose of ixazomib. Placebo Safety Population included all participants who received at least 1 dose of placebo. Adverse events are presented per treatment received during the course of the study.
Arm/Group | Ixazomib | Placebo
All-Cause Mortality (participants affected / at risk) | 1/35 | 0/4
Serious Adverse Events (participants affected / at risk) | 11/35 | 0/4
Other Adverse Events (participants affected / at risk) | 33/35 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib (N=35) | Placebo (N=4)
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib (N=35) | Placebo (N=4)
Anaemia (Blood and lymphatic system disorders) | 4 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Breath odour (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 12 | 1
Gastritis (Gastrointestinal disorders) | 2 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 6 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 9 | 0
Fatigue (General disorders) | 3 | 0
Peripheral swelling (General disorders) | 3 | 0
Pyrexia (General disorders) | 6 | 0
Hepatic steatosis (Hepatobiliary disorders) | 2 | 0
Bronchitis (Infections and infestations) | 4 | 0
COVID-19 (Infections and infestations) | 8 | 0
Herpes zoster (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 5 | 1
Pneumonia (Infections and infestations) | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 14 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 5 | 0
Neutrophil count decreased (Investigations) | 3 | 0
Platelet count decreased (Investigations) | 8 | 0
Weight decreased (Investigations) | 4 | 0
Weight increased (Investigations) | 2 | 1
White blood cell count decreased (Investigations) | 5 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 4 | 0
Headache (Nervous system disorders) | 4 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 0
Eczema (Skin and subcutaneous tissue disorders) | 4 | 0
Papule (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT03748953/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/53/NCT03748953/SAP_001.pdf